CLINICAL TRIAL: NCT01016977
Title: A Phase 4, Single-Blind, Randomized, Study to Compare the Tolerability and Efficacy of Tazorac Cream When Used in Combination With Either Duac Gel or Acanya Gel for the Treatment of Facial Acne Vulgaris
Brief Title: A Phase 4, Single-Blind, Randomized, Study to Compare the Tolerability and Efficacy of 0.1% Tazorac Cream When Used in Combination With Either Duac Gel or Acanya Gel for the Treatment of Facial Acne Vulgaris
Acronym: C0000-411
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 114566; NCT01334970 (obsolete NCT alias)
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Results first posted 2012-02-23 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin; Benzoyl Peroxide; tazarotene; clindamycin phosphate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duac & taz (Active Comparator): Clindamycin 1%/Benzoyl Peroxide 5% and 0.1% tazarotene
  Interventions: Drug: Clindamycin 1%/Benzoyl Peroxide 5% and 0.1% tazarotene
- Acanya & taz (Active Comparator): clindamycin phosphate 1.2%/benzoyl peroxide 2.5% and 0.1% tazarotene
  Interventions: Drug: clindamycin phosphate 1.2%/benzoyl peroxide 2.5% and 0.1% tazarotene

INTERVENTIONS:
Drug: Clindamycin 1%/Benzoyl Peroxide 5% and 0.1% tazarotene — Clindamycin 1%/Benzoyl Peroxide 5% and 0.1% tazarotene
  Arms: Duac & taz
Drug: clindamycin phosphate 1.2%/benzoyl peroxide 2.5% and 0.1% tazarotene — clindamycin phosphate 1.2%/benzoyl peroxide 2.5% and 0.1% tazarotene
  Arms: Acanya & taz

SUMMARY:
A single-blind (investigator-blinded), randomized, parallel group, single center study to evaluate the tolerability and efficacy of combination therapy with Duac Gel / 0.1% Tazorac Cream and Acanya Gel / 0.1% Tazorac Cream for the treatment of facial acne vulgaris.

DETAILED DESCRIPTION:
This is a single-blind (investigator-blinded), randomized, parallel group, single center study to evaluate the tolerability and efficacy of combination therapy with Duac Gel/Tazorac Cream and Acanya Gel/Tazorac Cream for the treatment of facial acne vulgaris. Approximately 40 male and female subjects will be enrolled (20 per study group).

Subjects will participate in the study for 12 weeks; visits will be scheduled at baseline and at weeks 1, 2, 4, 8, and 12 (total of 6 visits). Eligible subjects will be randomized at baseline to 1 of the 2 study groups in a 1:1 ratio (Duac Gel/Tazorac Cream to Acanya Gel/Tazorac Cream). Subjects will apply either Duac Gel or Acanya Gel to the face each morning and apply Tazorac Cream to the face each evening.

Tolerability will be evaluated through subject assessments of burning/stinging, itching, and oiliness and through investigator assessments of peeling, erythema, and dryness. In addition, subjects will evaluate their overall skin comfort and record the usage of moisturizer and sunscreen, if needed. Efficacy will be assessed through lesion counts (total, inflammatory and noninflammatory) and ISGA. Safety will be assessed by evaluating adverse events (AEs), concomitant medication use, and withdrawals from the study.

This is an investigator-blinded study; therefore, subjects and study-center staff will not be blinded to study treatment allocation. Subjects (and parents or legal guardians) and study-center staff will be instructed not to reveal study product allocation to the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of acne vulgaris.
* Lesion count: 20 to 50 inflammatory (papules and pustules) and 30 to 100 noninflammatory (open and closed - comedones) facial lesions excluding nose, and ≤ 1 small nodular lesion. Cystic lesions are not allowed at baseline.
* Investigator Static Global Assessment of 3 or 4 at Baseline.

Exclusion Criteria:

* Clinically relevant finding at baseline or medical history of severe systemic diseases or diseases of the facial skin, other than acne vulgaris.
* Subjects with cystic acne lesions.
* Facial hair that may obscure the accurate assessment of acne grade.
* History or presence of regional enteritis or inflammatory bowel disease (eg, ulcerative colitis, pseudomembranous colitis, chronic diarrhea, celiac disease or a history of antibiotic-associated colitis) or similar symptoms.
* Concurrent use of medications known to be photosensitizers (eg, thiazides, tetracyclines, fluoroquinolones, phenothiazines, and sulfonamides) because of the possibility of increased phototoxicity.
* Concomitant use of neuromuscular blocking agents. Clindamycin has neuromuscular blocking activities, which may enhance the action of other neuromuscular blocking agents.
* Use of topical anti-acne medications (eg, benzoyl peroxide, retinoids, azelaic acid, resorcinol, salicylates, sulfacetamide sodium and derivatives, and glycolic acid) within the past 2 weeks.
* Use of topical antibiotics on the face within the past 2 weeks or systemic antibiotics within the past 4 weeks.
* Use of topical corticosteroids on the face or systemic corticosteroids within the past 2 to 4 weeks, respectively. Use of inhaled, intra-articular or intra lesional (other than for facial acne lesions) steroids is acceptable.
* Use of systemic retinoids, such as Isotretinoin, within the past 6 months.
* Concomitant use of the following types of facial products: astringents, toners, abradants, hair removal wax, facials, peels containing glycolic or other acids, masks, washes or soaps containing benzoyl peroxide, sulfacetamide sodium or salicylic acid, non-mild facial cleansers, or moisturizers that contain retinol, salicylic acid, or α- or β hydroxy acids.
* Concomitant use of medications that are reported to exacerbate acne, (eg, vitamins such as vitamin D, vitamin A, vitamins B2, B6, B12; haloperidol, halogens such as iodide and bromide, lithium, cyclosporine, psoralen, sirolimus, imatinib, aripiprazole, isoniazid, valproate acid, hydantoin, and phenobarbital) as these may impact efficacy assessments. Iron supplements and folate are acceptable.
* Facial procedures (eg, chemical peel, lasers/lights, photodynamic therapy, microdermabrasion, artificial ultraviolet therapy) performed by an esthetician, beautician, physician, nurse, or other practitioner, within the past 4 weeks.
* Known hypersensitivity or previous allergic reaction to any component(s) or excipient(s) of the study products.
* Use of any investigational medications or treatments within the past 4 weeks.
* Treatment with estrogens, including oral, implanted and topical contraceptives, androgens, or anti-androgenic agents for 12 weeks or less immediately prior to starting study product and have not been prescribed for the treatment of Acne Vulgaris. Subjects that have been treated with estrogens, as described above, androgens, or anti androgenic agents for more than 12 consecutive weeks prior to start of study treatment are allowed to enroll as long as they do not expect to change dose, medication, or discontinue use during the study.
* Evidence of recent alcohol or drug abuse (in the opinion of the investigator).
* Live in the same household as currently enrolled subjects.
* Employee of the investigator, a clinical research organization, or Stiefel Laboratories who is involved in the study or an immediate family member (eg, partner, offspring, parents, siblings or sibling's offspring) of an employee involved in the study.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Dhawan SS, Gwazdauskas J. Clindamycin phosphate 1.2%-benzoyl peroxide (5% or 2.5%) plus tazarotene cream 0.1% for the treatment of acne. Cutis. 2013 Feb;91(2):99-104. PMID 23513559
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 114566 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114566 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114566 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114566 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114566 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114566 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114566 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Tazorac Cream/Duac Gel: Tazorac (tazarotene 0.1%) cream in evening (PM) and Duac (clindamycin 1%/benzoyl peroxide 5%) gel in morning (AM) daily for topical administration on face
- Tazorac Cream/Acanya Gel: Tazorac (tazarotene 0.1%) cream in PM and Acanya (clindamycin phosphate 1.2%/benzoyl peroxide 2.5%) gel in AM daily for topical administration on face
Period: Overall Study
Arm/Group | Tazorac Cream/Duac Gel | Tazorac Cream/Acanya Gel
Started | 20 | 20
Completed | 17 | 18
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tazorac Cream/Duac Gel | Tazorac Cream/Acanya Gel | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.2 (9.0) | 22.6 (7.8) | 21.9 (8.3)
Gender [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 7 | 11 | 18
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 8 | 15 | 23
  Black | 1 | 1 | 2
  White | 9 | 4 | 13
  Biracial, India, Black, and Phillipino | 1 | 0 | 1
  Multiracial (Black, White) | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Erythema at Weeks 1, 2, 4, 8, and 12
Description: Mean change from baseline was calculated as the average value at Weeks 1, 2, 4, 8, and 12 minus the value at baseline. Erythema (redness of the skin, due to increased blood flow in the capillaries in the lower layers of theh skin) was assessed by the investigator based on a 6-point scale: 0=none, which is normal; 1=trace, which is mild and localized; 2=mild, which is mild and diffuse; 3=moderate, which is moderate and diffuse; 4=marked, which is moderate and dense; 5=severe, which is prominent and dense.
Time Frame: Baseline and Weeks 1, 2, 4, 8, and 12
Population: Intent-to-Treat (ITT) Population: all randomized participants who received study product. Some participants did not return for all visits; thus, data were not captured for all participants in the ITT Population at all visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tazorac Cream/Duac Gel | Tazorac Cream/Acanya Gel
Number analyzed (Participants) | 20 | 20
units on a scale
  Week 1, n=19, 17 | 0.79 (1.03) | 0.76 (0.75)
  Week 2, n=20, 19 | 0.60 (0.82) | 0.47 (0.70)
  Week 4, n=20, 20 | 0.50 (0.89) | 0.55 (0.76)
  Week 8, n=20, 20 | 0.20 (0.62) | 0.20 (0.52)
  Week 12, n=20, 20 | 0.25 (0.64) | 0.10 (0.79)
Statistical Analysis 1: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.9597, ANCOVA — Week 1
Statistical Analysis 2: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.5538, ANCOVA — Week 2
Statistical Analysis 3: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.6315, ANCOVA — Week 4
Statistical Analysis 4: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.5655, ANCOVA — Week 8
Statistical Analysis 5: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.7917, ANCOVA — Week 12

2. Primary Outcome: Mean Change From Baseline in Dryness at Weeks 1, 2, 4, 8, and 12
Description: Mean change from baseline was calculated as the average value at Weeks 1, 2, 4, 8, and 12 minus the value at baseline. Dryness was assessed by the investigator based on a 6-point scale: 0=none, which is normal; 1=trace, which is mild and localized; 2=mild, which is mild and diffuse; 3=moderate, which is moderate and diffuse; 4=marked, which is moderate and dense; 5=severe, which is prominent and dense.
Time Frame: Baseline and Weeks 1, 2, 4, 8, and 12
Population: ITT Population. Some participants did not return for all visits; thus, data were not captured for all participants in the ITT Population at all visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tazorac Cream/Duac Gel: Tazorac (tazarotene 0.1%) cream in PM and Duac (clindamycin 1%/benzoyl peroxide 5%) gel in AM daily for topical administration on face
Arm/Group | Tazorac Cream/Duac Gel | Tazorac Cream/Acanya Gel
Number analyzed (Participants) | 20 | 20
units on a scale
  Week 1, n=19, 17 | 1.11 (1.05) | 1.18 (0.81)
  Week 2, n=20, 19 | 1.15 (0.81) | 0.84 (0.96)
  Week 4, n=20, 20 | 0.65 (0.75) | 0.55 (0.83)
  Week 8, n=20, 20 | 0.50 (0.95) | 0.15 (0.59)
  Week 12, n=20, 20 | 0.20 (0.70) | -0.05 (0.51)
Statistical Analysis 1: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.5961, ANCOVA — Week 1
Statistical Analysis 2: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.2293, ANCOVA — Week 2
Statistical Analysis 3: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.9852, ANCOVA — Week 4
Statistical Analysis 4: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.5538, ANCOVA — Week 8
Statistical Analysis 5: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.6540, ANCOVA — Week 12

3. Primary Outcome: Mean Change From Baseline in Peeling at Weeks 1, 2, 4, 8, and 12
Description: Mean change from baseline was calculated as the average value at Weeks 1, 2, 4, 8, and 12 minus the value at baseline. Peeling was assessed by the investigator based on a 6-point scale: 0=none, which is normal; 1=trace, which is mild and localized; 2=mild, which is mild and diffuse; 3=moderate, which is moderate and diffuse; 4=marked, which is moderate and dense; 5=severe, which is prominent and dense.
Time Frame: Baseline and Weeks 1, 2, 4, 8, and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tazorac Cream/Acanya Gel: Tazorac (tazarotene 0.1%) cream at PM and Acanya (clindamycin phosphate 1.2%/benzoyl peroxide 2.5%) gel in AM daily for topical administration on face
Arm/Group | Tazorac Cream/Duac Gel | Tazorac Cream/Acanya Gel
Number analyzed (Participants) | 20 | 20
units on a scale
  Week 1, n=19, 17 | 1.11 (1.05) | 1.06 (0.83)
  Week 2, n=20, 19 | 1.05 (0.83) | 0.79 (0.98)
  Week 4, n=20, 20 | 0.60 (0.75) | 0.55 (0.83)
  Week 8, n=20, 20 | 0.50 (0.95) | 0.10 (0.55)
  Week 12, n=20, 20 | 0.20 (0.70) | -0.05 (0.51)
Statistical Analysis 1: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.8545, ANCOVA — Week 1
Statistical Analysis 2: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.2895, ANCOVA — Week 2
Statistical Analysis 3: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.8234, ANCOVA — Week 4
Statistical Analysis 4: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.3644, ANCOVA — Week 8
Statistical Analysis 5: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.6540, ANCOVA — Week 12

4. Primary Outcome: Mean Change From Baseline in Burning/Stinging at Weeks 1, 2, 4, 8, and 12
Description: Mean change from baseline was calculated as the average value at Weeks 1, 2, 4, 8, and 12 minus the value at baseline. Burning/stinging was assessed by participants based on a 6-point scale: 0=none: normal, no discomfort; 1=trace: awareness, no discomfort, no intervention required; 2=mild: noticeable discomfort, intermittent awareness; 3=moderate: noticeable discomfort, continuous awareness; 4=marked: definite discomfort, continuous awareness, interferes occasionally with normal daily activities; 5=severe: definite continuous discomfort, interferes with normal daily activities.
Time Frame: Baseline and Weeks 1, 2, 4, 8, and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tazorac Cream/Duac Gel | Tazorac Cream/Acanya Gel
Number analyzed (Participants) | 20 | 20
units on a scale
  Week 1, n=19, 17 | 1.58 (1.87) | 1.65 (1.69)
  Week 2, n=20, 19 | 0.70 (1.59) | 0.84 (1.07)
  Week 4, n=20, 20 | 1.25 (1.92) | 0.55 (0.76)
  Week 8, n=20, 20 | 0.60 (1.27) | 0.45 (0.69)
  Week 12, n=20, 20 | 0.50 (1.40) | 0.40 (0.82)
Statistical Analysis 1: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.7546, ANCOVA — Week 1
Statistical Analysis 2: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.7705, ANCOVA — Week 2
Statistical Analysis 3: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.0259, ANCOVA — Week 4
Statistical Analysis 4: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.9252, ANCOVA — Week 8
Statistical Analysis 5: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.2927, ANCOVA — Week 12

5. Primary Outcome: Mean Change From Baseline in Itching at Weeks 1, 2, 4, 8, and 12
Description: Mean change from baseline was calculated as the average value at Weeks 1, 2, 4, 6, 8, and 12 minus the value at baseline. Itching was assessed by participants based on a 6-point scale: 0=none: normal, no discomfort; 1=trace: awareness, no discomfort, no intervention required; 2=mild: noticeable discomfort, intermittent awareness; 3=moderate: noticeable discomfort, continuous awareness; 4=marked: definite discomfort, continuous awareness, interferes occasionally with normal daily activities; 5=severe: definite continuous discomfort, interferes with normal daily activities.
Time Frame: Baseline and Weeks 1, 2, 4, 8, and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tazorac Cream/Duac Gel | Tazorac Cream/Acanya Gel
Number analyzed (Participants) | 20 | 20
units on a scale
  Week 1, n=19, 17 | 0.68 (1.57) | 0.76 (1.64)
  Week 2, n=20, 19 | 0.10 (0.79) | 0.84 (1.38)
  Week 4, n=20, 20 | 0.20 (1.20) | 0.65 (1.18)
  Week 8, n=20, 20 | -0.05 (1.15) | 0.30 (0.80)
  Week 12, n=20, 20 | 0.35 (1.42) | 0.45 (1.47)
Statistical Analysis 1: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.4010, ANCOVA — Week 1
Statistical Analysis 2: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.0963, ANCOVA — Week 2
Statistical Analysis 3: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.9291, ANCOVA — Week 4
Statistical Analysis 4: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.5523, ANCOVA — Week 8
Statistical Analysis 5: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.2556, ANCOVA — Week 12

6. Primary Outcome: Mean Change From Baseline in Oiliness at Weeks 1, 2, 4, 8, and 12
Description: Mean change from baseline was calculated as the average value at Weeks 1, 2, 4, 8, and 12 minus the value at baseline. Oiliness was assessed by participants based on a 6-point scale: 0=none: normal, no discomfort; 1=trace: awareness, no discomfort, no intervention required; 2=mild: noticeable discomfort, intermittent awareness; 3=moderate: noticeable discomfort, continuous awareness; 4=marked: definite discomfort, continuous awareness, interferes occasionally with normal daily activities; 5=severe: definite continuous discomfort, interferes with normal daily activities.
Time Frame: Baseline and Weeks 1, 2, 4, 8, and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tazorac Cream/Duac Gel | Tazorac Cream/Acanya Gel
Number analyzed (Participants) | 20 | 20
units on a scale
  Week 1, n=19, 17 | -1.00 (1.60) | -1.29 (1.40)
  Week 2, n=20, 19 | -0.95 (1.61) | -1.05 (1.35)
  Week 4, n=20, 20 | -0.85 (1.87) | -0.55 (1.85)
  Week 8, n=20, 20 | -0.80 (1.79) | -1.05 (1.39)
  Week 12, n=20, 20 | -0.35 (1.84) | -0.75 (1.97)
Statistical Analysis 1: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.4037, ANCOVA — Week 1
Statistical Analysis 2: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.8662, ANCOVA — Week 2
Statistical Analysis 3: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.5951, ANCOVA — Week 4
Statistical Analysis 4: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.2349, ANCOVA — Week 8
Statistical Analysis 5: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.3461, ANCOVA — Week 12

7. Primary Outcome: Mean Change From Baseline in Skin Overall Comfort at Weeks 1, 2, 4, 8, and 12
Description: Mean change from baseline was calculated as the average value at Weeks 1, 2, 4, 8, and 12 minus the value at baseline. Skin comfort was assessed by participants based on 5-point scale: +2, very comfortable; +1, comfortable; 0, neutral; -1, somewhat uncomfortable; or -2, uncomfortable.
Time Frame: Baseline and Weeks 1, 2, 4, 8, and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tazorac Cream/Duac Gel | Tazorac Cream/Acanya Gel
Number analyzed (Participants) | 20 | 20
units on a scale
  Week 1, n=19, 17 | -0.37 (1.54) | -0.29 (0.92)
  Week 2, n=20, 19 | 0.25 (1.45) | 0.05 (0.91)
  Week 4, n=20, 20 | 0.05 (1.23) | -0.10 (0.85)
  Week 8, n=20, 20 | 0.30 (1.17) | 0.10 (0.85)
  Week 12, n=20, 20 | 0.45 (1.39) | 0.60 (0.99)
Statistical Analysis 1: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.7250, ANCOVA — Week 1
Statistical Analysis 2: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.9743, ANCOVA — Week 2
Statistical Analysis 3: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.9816, ANCOVA — Week 4
Statistical Analysis 4: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.8809, ANCOVA — Week 8
Statistical Analysis 5: Comparison: Tazorac Cream/Duac Gel vs Tazorac Cream/Acanya Gel; Test type: Superiority or Other; p = 0.1679, ANCOVA — Week 12

8. Secondary Outcome: Number of Participants With at Least a Two-grade Improvement in ISGA Score From Baseline to Week 12
Description: The investigator conducted the overall assessment of the participant's facial acne vulgaris based on the Investigator's Static Global Assessment Scale (ISGA). The ISGA is a 6-point scale: 0, clear skin with no acne vulgaris; 1, almost clear skin; 2, mild; 3, moderate; 4, severe; 5, very severe.
Time Frame: Baseline and Week 12
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Tazorac Cream/Duac Gel | Tazorac Cream/Acanya Gel
Number analyzed (Participants) | 20 | 20
participants | 7 | 10

9. Secondary Outcome: Mean Change From Baseline in Inflammatory and Non-inflammatory Lesion Counts at Weeks 1, 2, 4, 8, and 12
Description: Inflammation is defined as a localized protective reaction of tissue to irritation, injury, or infection, characterized by pain, redness, swelling, and sometimes loss of function. The investigator counted inflammatory (papules, pustules, and nodules) and non-inflammatory (open and closed comedones) lesions on a participant's face at each study visit. The face is defined as the hairline edge to the mandibular line and should include the forehead, cheeks, and chin. W, Week.
Time Frame: Baseline and Weeks 1, 2, 4, 8, and 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Tazorac Cream/Duac Gel | Tazorac Cream/Acanya Gel
Number analyzed (Participants) | 20 | 20
lesions
  W1, Inflammatory lesions, n=19, 17 | -6.6 (5.3) | -5.9 (6.1)
  W2, Inflammatory lesions, n=20, 19 | -8.8 (8.7) | -8.1 (6.3)
  W4, Inflammatory lesions, n=20, 20 | -13.0 (6.3) | -9.6 (9.2)
  W8, Inflammatory lesions, n=20, 20 | -14.9 (7.2) | -16.3 (5.7)
  W12, Inflammatory lesions, n=20, 20 | -18.0 (6.6) | -13.4 (13.6)
  W1, Non-inflammatory lesions, n=19, 17 | -3.2 (11.2) | -7.6 (7.1)
  W2, Non-inflammatory lesions, n=20, 19 | -17.9 (11.4) | -15.1 (11.4)
  W4, Non-inflammatory lesions, n=20, 20 | -23.6 (13.6) | -26.6 (13.2)
  W8, Non-inflammatory lesions, n=20, 20 | -28.9 (19.1) | -33.1 (17.3)
  W12, Non-inflammatory lesions, n=20, 20 | -32.6 (19.4) | -37.8 (21.4)

10. Secondary Outcome: Mean Change From Baseline in Total Lesion Count at Weeks 1, 2, 4, 8, and 12
Description: The investigator will count inflammatory (papules, pustules, and nodules) and non-inflammatory (open and closed comedones) lesions on the participant's face at each study visit. The face is defined as the hairline edge to the mandibular line and should include the forehead, cheeks, and chin.
Time Frame: Baseline and Weeks 1, 2, 4, 8, and 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Tazorac Cream/Duac Gel | Tazorac Cream/Acanya Gel
Number analyzed (Participants) | 20 | 20
lesions
  Week 1, n=19, 17 | -9.8 (14.0) | -13.5 (9.4)
  Week 2, n=20, 19 | -26.6 (15.3) | -23.1 (14.5)
  Week 4, n=20, 20 | -36.6 (15.4) | -36.2 (15.4)
  Week 8, n=20, 20 | -43.7 (23.5) | -49.4 (20.2)
  Week 12, n=20, 20 | -50.6 (23.1) | -51.1 (27.8)

11. Secondary Outcome: Mean Change From Baseline for the Global Score of the Participant-completed Skindex-29 Quality of Life Questionnaire at Week 12
Description: Skindex-29 is a 3-component (symptomatic, emotional, and functional) self-administered questionnaire (comprised of 30 questions) used to comprehensively measure the complex effects of skin diseases on a participant's quality of life. Participants were asked to answer questions based on a 5-point scale concerning their feelings over the past 4 weeks about the skin condition that has bothered them the most: 1, never; 2, rarely; 3, sometimes; 4, often; 5, all the time. The Global Score is the sum of the 30 question scores; total score ranges from 30 to 150.
Time Frame: Baseline and Week 12
Population: ITT Population. Participants with missing baseline values were not included in this analysis. No sunscreen or moisturizer data were collected; thus, there was no analysis of these data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tazorac Cream/Acanya Gel: Tazorac cream in PM and Acanya (clindamycin phosphate 1.2%/benzoyl peroxide 2.5%) gel in AM daily for topical administration on face
Arm/Group | Tazorac Cream/Duac Gel | Tazorac Cream/Acanya Gel
Number analyzed (Participants) | 18 | 19
units on a scale | -6.1 (11.6) | -3.7 (8.4)

12. Secondary Outcome: Mean Change From Baseline for the Symptomatic Score of the Participant-completed Skindex-29 Quality of Life Questionnaire at Week 12
Description: Skindex-29 is a 3-component (symptomatic, emotional, and functional) self-administered questionnaire (comprised of 30 questions) used to comprehensively measure the complex effects of skin diseases on a participant's quality of life. Participants were asked to answer questions based on a 5-point scale concerning their feelings over the past 4 weeks about the skin condition that has bothered them the most: 1, never; 2, rarely; 3, sometimes; 4, often; 5, all the time. The Symptomatic Score is the sum of 7 question scores; total score ranges from 7 to 35.
Time Frame: Baseline and Week 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tazorac Cream/Duac Gel | Tazorac Cream/Acanya Gel
Number analyzed (Participants) | 18 | 19
units on a scale | -8.7 (15.7) | -1.4 (13.5)

13. Secondary Outcome: Mean Change From Baseline for the Emotional Score of the Participant-completed Skindex-29 Quality of Life Questionnaire at Week 12
Description: Skindex-29 is a 3-component (symptomatic, emotional, and functional) self-administered questionnaire (comprised of 30 questions) used to comprehensively measure the complex effects of skin diseases on a participant's quality of life. Participants were asked to answer questions based on a 5-point scale concerning their feelings over the past 4 weeks about the skin condition that has bothered them the most: 1, never; 2, rarely; 3, sometimes; 4, often; 5, all the time. The Emotional Score is the sum of 10 question scores; total score ranges from 10 to 50.
Time Frame: Baseline and Week 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tazorac Cream/Duac Gel | Tazorac Cream/Acanya Gel
Number analyzed (Participants) | 18 | 19
units on a scale | -11.2 (11.8) | -7.1 (8.9)

14. Secondary Outcome: Mean Change From Baseline for the Functional Score of the Participant-completed Skindex-29 Quality of Life Questionnaire at Week 12
Description: Skindex-29 is a 3-component (symptomatic, emotional, and functional) self-administered questionnaire (comprised of 30 questions) used to comprehensively measure the complex effects of skin diseases on a participant's quality of life. Participants were asked to answer questions based on a 5-point scale concerning their feelings over the past 4 weeks about the skin condition that has bothered them the most: 1, never; 2, rarely; 3, sometimes; 4, often; 5, all the time. The Functional Score is the sum of 12 question scores; total score ranges from 12 to 60.
Time Frame: Baseline and Week 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tazorac Cream/Duac Gel | Tazorac Cream/Acanya Gel
Number analyzed (Participants) | 18 | 19
units on a scale | -6.1 (11.6) | -3.7 (8.4)

15. Secondary Outcome: Overall Satisfaction With Study Product at Week 12
Description: Overall satisfaction with the study product was assessed from a participant's answer to the following question on the product acceptability and preference questionnaire at the end of study (i.e., Week 12): "What is your overall satisfaction with the study product." Participants assessed overall satisfaction with the study product in the morning and evening, based on a 6-point scale: 1, very satisfied; 2, satisfied; 3, neutral (no opinion); 4, unsatisfied; 5, very unsatisfied.
Time Frame: Week 12
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tazorac Cream/Duac Gel | Tazorac Cream/Acanya Gel
Number analyzed (Participants) | 20 | 20
units on a scale
  Morning | 1.76 (1.15) | 1.75 (0.72)
  Evening | 1.59 (1.00) | 1.70 (0.92)

ADVERSE EVENTS:
Arm/Group | Tazorac Cream/Duac Gel | Tazorac Cream/Acanya Gel
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 11/20 | 7/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tazorac Cream/Duac Gel (N=20) | Tazorac Cream/Acanya Gel (N=20)
Nasopharyngitis (Infections and infestations) | 6 | 6
Bacterial Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Viral Infection (Infections and infestations) | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Application Site Erythema (General disorders) | 1 | 0
Application Site Irritation (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.